CLINICAL TRIAL: NCT00718861
Title: A 3-year, Multicenter, Double-blind, Randomized, Placebo-controlled Extension to CZOL446H2301E1 to Evaluate the Efficacy and Long Term Safety of 6 and 9 Years Zoledronic Acid Treatment of Postmenopausal Women With Osteoporosis
Brief Title: 3 yr Efficacy & Safety Study of Zoledronic Acid in Post-menopausal Women With Osteoporosis Treated With Zol Acid for 6 Yrs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446H2301E2; 2007-005383-27 (EudraCT Number)
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-09

CONDITIONS: Post-menopausal Osteoporosis
Keywords: Osteoporosis; zoledronic acid; post-menopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo administered intravenously.
  Interventions: Drug: Placebo
- Zoledronic acid (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Zoledronic acid
  Other Names: Reclast®, Aclasta®
  Arms: Zoledronic acid

SUMMARY:
This second extension will evaluate the efficacy and long term safety of zoledronic acid in women with post-menopausal osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* Women who have received the 4th and 6th dose of zoledronic acid in study CZOL446H2301E1

Exclusion Criteria:

* Poor kidney, eye, liver health
* Use of certain therapies for osteoporosis in study CZOL446H2301E1
* Abnormal calcium levels

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (10):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Lakewood, Colorado
  - Novartis Investigative Site, Gainesville, Georgia
  - Novartis Investigative Site, Indiamapolis, Indiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Seattle, Washington
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
- Australia (3):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Colombia (3):
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
- Novartis Investigative Site, Helsinki, Finland
- Novartis Investigative Site, Lyon, France, France
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Braunfels
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (4):
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Győr
- Italy (4):
  - Novartis Investigative Site, Arenzano, GE
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Valeggio sul Mincio, VR
- Novartis Investigative Site, Grafton, Auckland, New Zealand
- Norway (3):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Hamar
  - Novartis Investigative Site, Oslo
- Poland (3):
  - Novartis Investigative Site, Warsaw, Poland
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Warsaw
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Thailand (2):
  - Novartis Investigative Site, Chaingmai
  - Novartis Investigative Site, Khonkaen

RESULTS

PARTICIPANT FLOW:
Groups:
- Z9 (Zoledronic Acid 9): Group Z9 patients were those who had been treated with zoledronic acid for up to 9 years in the core (CZOL446H2301) and extension studies (CZOL446H2301E1 and CZOL446H2301E2).
- Z6P3 (Zoledronic Acid 6 Placebo 3): Group Z6P3 patients were those who had been treated with zoledronic acid for 6 years in the core (CZOL446H2301) and the first extension study (CZOL446H2301E1) followed by up to 3 years of placebo in the second extension study (CZOL446H2301E2).
Period: Overall Study
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Started | 95 ("Started" indicates Randomized and Intent-to Treat (ITT) population) | 95
Safety Set | 92 (3 patients randomized but never received study drug) | 95
Modified Intent to Treat | 67 (ITT patients with DXA total hip measure at extension 2 baseline and year 9) | 69 (ITT patients with DXA total hip measure at extension 2 baseline and year 9)
Completed | 74 | 77
Not Completed | 21 | 18
Not completed — Withdrawal by Subject | 15 | 10
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Administrative Problems | 1 | 1
Not completed — Death | 1 | 5

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all patients who were enrolled in the extension study at Visit 12. This included patients who were randomized to Z9 and Z6P3 groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3) | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78 (4.71) | 78.1 (4.85) | 78.1 (4.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 95 | 190
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Total Hip Bone Mineral Density BMD at Year 6 (Baseline) and Year 9
Description: Bone Mineral Density (BMD) measured by dual energy x-ray absorptiometry (DXA). DXA consists of two X-ray beams with different energy levels that are aimed at the patient's bones. When soft tissue absorption is subtracted out, the BMD can be determined from the absorption of each beam by bone. Percentage change from Year 6 = 100*(Year 9 - Year 6)/Year 6.
Time Frame: Year 6 (baseline) and Year 9
Population: The modified intent-to-treat (MITT) population included all patients in the ITT population who had DXA measurements of the total hip at Visit 11 (Year 6) and Visit 15 (Year 9). This was the primary population for the primary efficacy parameter.
Measure: Least Squares Mean (Standard Error); unit: Percentage Change of BMD
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 67 | 69
Percentage Change of BMD | -0.54 (0.433) | -1.31 (0.427)

2. Secondary Outcome: Percentage Change of Total Hip Bone Mineral Density (BMD) at Year 7 and 8 Compared to Year 6
Description: as for outcome 1
Time Frame: Year 6 (extension 2 baseline), Year 7, Year 8
Population: The intent-to-treat (ITT) population included all patients who were enrolled in the extension study at Visit 12. This included patients who were randomized to Z9 and Z6P3 groups. n = the number of patients with measurements at Year 6 and follow-up visits as determined by the analysis window.
Measure: Least Squares Mean (Standard Error); unit: percentage change of BMD
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
percentage change of BMD
  Year 7 (n=83,76) | -0.28 (0.336) | -0.83 (0.347)
  Year 8 (n=73,72) | -0.14 (0.311) | -1.06 (0.315)

3. Secondary Outcome: Percentage Change of Femoral Neck Bone Mineral Density (BMD) at Year 7, 8 and 9 Compared to Year 6
Description: as for outcome 1
Time Frame: Year 6 (extension 2 baseline), Year 7, Year 8, Year 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change of BMD
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
percentage change of BMD
  Year 7 (n=83,76) | -0.78 (0.433) | -1.24 (0.447)
  Year 8 (n=73,72) | 0.00 (0.521) | -0.88 (0.528)
  Year 9 (n=67,69) | -1.11 (0.554) | -1.17 (0.547)

4. Secondary Outcome: Percentage Change of Total Hip Bone Mineral Density (BMD) at Year 7, 8 and 9 Compared to Year 0
Description: Bone Mineral Density (BMD) measured by dual energy x-ray absorptiometry (DXA). DXA consists of two X-ray beams with different energy levels that are aimed at the patient's bones. When soft tissue absorption is subtracted out, the BMD can be determined from the absorption of each beam by bone. Percentage change from Year 0 = 100*(Year 9 - Year 0)/Year 0.
Time Frame: Year 0 (core baseline), Year 7, Year 8, Year 9
Population: The intent-to-treat (ITT) population included all patients who were enrolled in the extension study at Visit 12. This included patients who were randomized to Z9 and Z6P3 groups. n = the number of patients with measurements at Year 0 and follow-up visits as determined by the analysis window.
Measure: Least Squares Mean (Standard Error); unit: percentage change of BMD
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
percentage change of BMD
  Year 7 (n=83,75) | 4.81 (0.619) | 3.73 (0.640)
  Year 8 (n=72,71) | 5.35 (0.677) | 3.65 (0.684)
  Year 9 (n=67,68) | 4.64 (0.760) | 3.68 (0.752)

5. Secondary Outcome: Percentage Change of Femoral Neck Bone Mineral Density (BMD) at Year 7, 8 and 9 Compared to Year 0
Description: as for outcome 4
Time Frame: Year 0 (core baseline), Year 7, Year 8, Year 9
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage change of BMD
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
percentage change of BMD
  Year 7 (n=83,75) | 5.11 (0.921) | 3.86 (0.952)
  Year 8 (n=72,71) | 6.12 (1.041) | 4.43 (1.052)
  Year 9 (n=67,68) | 4.16 (0.963) | 3.88 (0.954)

6. Secondary Outcome: Biomarkers (Bone Markers) Serum C-terminal Telopeptide of Type I Collagen (CTx) at Year 6 (Extension 2 Baseline), Year 7, Year 8, Year 9
Description: Bone marker analysis: All patients had blood samples collected for analysis of serum c-terminal telopeptide of type I collagen (CTx). Serum CTX assays measure a fragment of the C-terminal telopeptide of type 1 collagen released during resorption of mature bone
Time Frame: Year 6 (extension 2 baseline), Year 7, Year 8, Year 9
Population: The intent-to-treat (ITT) population included all patients who were enrolled in the extension study at Visit 12. This included patients who were randomized to Z9 and Z6P3 groups. n = the number of patients with measurements at each visit as determined by the analysis window.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
ng/ml
  Year 6 (n=59, 58) | 0.19 [0.1 to 0.6] | 0.18 [0.1 to 0.5]
  Year 7 (n=56, 51) | 0.2 [0.1 to 0.4] | 0.22 [0.1 to 0.5]
  Year 8 (n=51, 52) | 0.22 [0.1 to 0.4] | 0.2 [0.1 to 0.4]
  Year 9 (n=51,54) | 0.22 [0.1 to 0.6] | 0.22 [0.1 to 0.7]

7. Secondary Outcome: Biomarkers (Bone Markers)Serum N-terminal Propeptide of Type I Collagen (P1NP) at Year 6 (Extension 2 Baseline), Year 7, Year 8, Year 9
Description: Bone marker analysis: All patients had blood samples collected for analysis of serum n-terminal propeptide of type I collagen (P1NP) The P1NP concentration is directly proportional to the amount of new collagen laid down during bone formation.
Time Frame: Year 6 (extension 2 baseline), Year 7, Year 8, Year 9
Population: as for outcome 6
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
ng/ml
  Year 6 (n=88, 86) | 25.89 [10.8 to 69.1] | 24.98 [9.9 to 65.6]
  Year 7 (n=58, 65) | 25.69 [12.3 to 52.9] | 27.79 [11.7 to 140.2]
  Year 8 (n=54, 57) | 26.07 [10.9 to 59.9] | 25.19 [13.1 to 68.1]
  Year 9 (n=52,56) | 26.74 [12.4 to 133.4] | 27.41 [11.3 to 119.4]

8. Secondary Outcome: Biomarkers (Bone Markers) Serum Bone-specific Alkaline Phosphatase (BSAP). at Year 6 (Extension 2 Baseline), Year 7, Year 8, Year 9
Description: Bone marker analysis: All patients had blood samples collected for analysis of serum bone-specific alkaline phosphatase (BSAP).Bone-specific alkaline phosphatase (BSAP) is a useful marker of active bone formation.
Time Frame: Year 6 (extension 2 baseline), Year 7, Year 8, Year 9
Population: as for outcome 6
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
ng/ml
  Year 6 (n=59, 62) | 8.16 [4.9 to 15.9] | 8.95 [3.9 to 16.2]
  Year 7 (n=58, 65) | 8.4 [4.7 to 15.7] | 10.00 [5.1 to 19.6]
  Year 8 (n=54, 57) | 7.84 [5.4 to 16.4] | 9.57 [5.6 to 15.8]
  Year 9 (n=52, 56) | 8.46 [5.1 to 18.3] | 9.94 [6.2 to 20.7]

9. Secondary Outcome: Number of Participants With New/Worsening Morphometric Vertebral Fractures at Year 9 Compared to Year 6
Description: Morphometric vertebral fracture (VF) was assessed based on morphometry. QM (quantitative morphometry) incident VF(QM positive) was defined by at least a 20% decrease in any vertebral height (at least 4 mm). If a participant had a QM positive at any vertebrae at any visit, x-rays from all visits for participants were evaluated using Genant semi-quantitative (SQ) method for VF assessment. A fracture was defined as an SQ reading that was greater than the baseline SQ reading.
Time Frame: Year 6 (extension 2 baseline), Year 9 (3 years of study duration)
Population: The intent-to-treat (ITT) population included all patients who were enrolled in the extension study at Visit 12. This included patients who were randomized to Z9 and Z6P3 groups. n= the number of patients with the event
Measure: Number; unit: participants
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
participants
  New Morphometric vertebral fracture | 3 | 5
  New/worsening Morphometric vertebra | 3 | 5

10. Secondary Outcome: Mean of Time to First Clinical Fracture
Description: The mean of time to the first clinical fracture is estimated from the area under the Kaplan-Meier curve.
Time Frame: over 3 years of study duration
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Days
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
Days | 1212.05 (22.96) | 1204.65 (26.35)

11. Secondary Outcome: Change in Height at Years 7, 8 and 9 Relative to Year 6
Description: Height was measured using a stadiometer in millimeters (mm). A stadiometer is a piece of medical equipment used for measuring height. It is usually constructed out of a ruler and a sliding horizontal headpiece which is adjusted to rest on the top of the head.
Time Frame: Year 6 (extension 2 baseline), Year 7, Year 8, Year 9
Population: The intent-to-treat (ITT) population included all patients who were enrolled in the extension study at Visit 12. This included patients who were randomized to Z9 and Z6P3 groups. n = the number of patients with evaluable measurements at both Year 6 and the post-Year 6 visit, as determined by the analysis window.
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Number analyzed (Participants) | 95 | 95
millimeters (mm)
  Year 7 (n=58, 51) | -5.29 (1.171) | -4.84 (1.199)
  Year 8 (n=55, 49) | -10.16 (1.875) | -9.90 (2.006)
  Year 9 (n=52, 48) | -13.31 (1.975) | -11.65 (2.085)

ADVERSE EVENTS:
Description: The safety population included all patients in the Intent to Treat (ITT) population who received at least 1 dose of study drug during this second extension study. Adverse Events data used the safety population.
Arm/Group | Z9 (Zoledronic Acid 9) | Z6P3 (Zoledronic Acid 6 Placebo 3)
Serious Adverse Events (participants affected / at risk) | 24/92 | 28/95
Other Adverse Events (participants affected / at risk) | 62/92 | 58/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Z9 (Zoledronic Acid 9) (N=92) | Z6P3 (Zoledronic Acid 6 Placebo 3) (N=95)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Oesophageal discomfort (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Z9 (Zoledronic Acid 9) (N=92) | Z6P3 (Zoledronic Acid 6 Placebo 3) (N=95)
Atrial fibrillation (Cardiac disorders) | 5 | 1
Cataract (Eye disorders) | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Fatigue (General disorders) | 5 | 2
Bronchitis (Infections and infestations) | 5 | 9
Cystitis (Infections and infestations) | 5 | 5
Nasopharyngitis (Infections and infestations) | 9 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 10 | 8
Contusion (Injury, poisoning and procedural complications) | 2 | 7
Fall (Injury, poisoning and procedural complications) | 8 | 11
Creatinine renal clearance decreased (Investigations) | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 1
Sciatica (Nervous system disorders) | 1 | 5
Insomnia (Psychiatric disorders) | 5 | 1
Hypertension (Vascular disorders) | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.